CLINICAL TRIAL: NCT02626026
Title: A Phase 1, Placebo-Controlled, Randomized Study Evaluating the Safety and Pharmacokinetics of GS-4059 in Healthy Volunteers and Subjects With Rheumatoid Arthritis (RA)
Brief Title: Study to Evaluate Safety and Pharmacokinetics of GS-4059 (Tirabrutinib) in Healthy Volunteers and Participants With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-407-1833; 2015-003240-40 (EudraCT Number)
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tirabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1, Part A: Tirabrutinib 20 mg QD (Experimental): Tirabrutinib 20 mg capsules orally once daily (QD) in the morning for 1 week.
  Interventions: Drug: Tirabrutinib
- Cohort 1, Part A: Placebo (Placebo Comparator): Placebo to match tirabrutinib capsules orally QD in the morning for 1 week.
  Interventions: Drug: Placebo
- Cohort 2, Part A: Tirabrutinib 10 mg BID (Experimental): Tirabrutinib 10 mg capsules orally twice daily (BID) (morning and approximately 12 hours later) for 7 days. On Day 7, only morning dose was administered.
  Interventions: Drug: Tirabrutinib
- Cohort 2, Part A: Placebo (Placebo Comparator): Placebo to match tirabrutinib capsules orally BID (morning and approximately 12 hours later) for 7 days. On Day 7, only morning dose was administered.
  Interventions: Drug: Placebo
- Part B: Tirabrutinib 20 mg QD (Experimental): Tirabrutinib 20 mg capsules orally QD for 4 weeks.
  Interventions: Drug: Tirabrutinib
- Part B: Placebo (Placebo Comparator): Placebo to match tirabrutinib capsules orally QD for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirabrutinib — Capsules administered orally.
  Other Names: GS-4059
  Arms: Cohort 1, Part A: Tirabrutinib 20 mg QD; Cohort 2, Part A: Tirabrutinib 10 mg BID; Part B: Tirabrutinib 20 mg QD
Drug: Placebo — Capsules administered orally.
  Arms: Cohort 1, Part A: Placebo; Cohort 2, Part A: Placebo; Part B: Placebo

SUMMARY:
This study will consist of two parts: Part A will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of tirabrutinib in healthy participants. Part B will evaluate the safety, tolerability, and the effect of tirabrutinib on disease-specific clinical markers and outcomes in participants with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria

Part A

* Be a nonsmoker
* Have a calculated body mass index (BMI) from 19 to 30 kg/m^2, inclusive, at screening
* Have a creatinine clearance (CrCl) ≥ 90 mL/min (using the Cockcroft-Gault method based on serum creatinine and actual body weight as measured at screening
* Females of childbearing potential must have a negative serum pregnancy test at screening and clinic admission.
* Male and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Must, in the opinion of the investigator, be in good health based upon medical history and physical examination, including vital signs
* Screening laboratory evaluations (hematology including reticulocytes, fasting lipids, chemistry, and urinalysis) must fall within the normal range of the local laboratory's reference ranges unless the results have been determined by the investigator to have no clinical significance
* Have either a normal 12-lead ECG or one with abnormalities that are considered clinically insignificant by the investigator in consultation with the Sponsor

Part B

* Diagnosis of RA (according to the 1987 American College of Rheumatology (ACR) classification criteria OR a score of ≥ 6 as defined by the ACR/European League Against Rheumatism Classification and Diagnostic Criteria for RA)
* Individuals must have taken methotrexate (MTX) 7.5 to 25 mg/week continuously for at least 12 weeks, with at least 6 weeks of stable dose prior to first study drug dose and throughout study duration.
* Individuals must be receiving folic or folinic acid supplementation at a stable dose for at least 6 weeks prior to Day 1 dosing and throughout study duration
* Individuals are allowed to remain on anti-malarial therapy, with at least 8 weeks of stable dose prior to first study drug dose
* Use of oral corticosteroids of no more than 10 mg prednisone or its equivalent per day is allowed if dose is stable for at least 28 days prior to first study drug dose
* Nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesics (including aspirin ≤ 100 mg daily) are allowed if doses are stable for at least 14 days prior to the first dose of study drug
* Estimated creatinine clearance (CLCr) ≥ 60 mL/min (using the Cockcroft-Gault method) based on serum creatinine and actual body weight as measured at the screening evaluation
* White blood cells (WBC), neutrophil count, lymphocyte count, and platelet count ≥ 0.75 x lower limit of normal (LLN)
* A negative serum pregnancy test at screening and a negative pregnancy test on the Day 1 visit prior to the first dose of study drug for female individual of child bearing potential.
* Male and female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Exclusion Criteria

Part A

* Pregnant or lactating individuals
* Have any serious or active medical or psychiatric illness (including depression) which, in the opinion of the Investigator, would interfere with individual's treatment, assessment, or compliance with the protocol. This would include renal, cardiac, hematological, hepatic, pulmonary (including chronic asthma), endocrine (including diabetes), central nervous, gastrointestinal (including an ulcer), vascular, metabolic (thyroid disorders, adrenal disease), immunodeficiency disorders, active infection, or malignancy that are clinically significant or requiring treatment
* Positive test for drugs of abuse, including alcohol at screening or on Day -1/check-in
* A positive test result for human immunodeficiency virus (HIV-1) antibody, hepatitis B (HBV) surface antigen or hepatitis C (HCV) antibody
* Have poor venous access that limits phlebotomy
* Have taken any prescription medications or over-the-counter medications, including herbal products, within 28 days prior to start of study drug dosing, with the exception of vitamins and/or acetaminophen and/or hormonal contraceptive medications
* Have been treated with systemic steroids, immunosuppressant therapies, or chemotherapeutic agents within 3 months prior to Screening or expected to receive these agents during the study (eg, corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies)
* Significant drug sensitivity or drug allergy (such as anaphylaxis or hepatoxicity)
* Medical or surgical treatment that permanently alters gastric absorption (eg, gastric or intestinal surgery); a history of cholecystectomy is not exclusionary

Part B

* Known hypersensitivity to formulation excipient.
* Pregnant or lactating females
* Previous treatment with B-cell depleting agents (eg, rituximab) within 12 months of treatment
* Prior treatment with any commercially available or investigational Bruton's tyrosine kinase (BTK) inhibitor
* Diagnosis of diabetes, history of impaired glucose tolerance test, history of abnormal glycated haemoglobin (HbA1c), or history of impaired fasting glucose
* Current treatment with any other disease modifying anti-rheumatic drug (DMARD) other than MTX and hydroxychloroquine, unless appropriate wash out
* Current treatment with any biologic agent, unless appropriate wash out
* Any laboratory abnormality or condition that, in the investigator's opinion, could adversely affect the safety of the individual or impair the assessment of study results
* History of or current inflammatory joint disease, other than RA
* Active significant systemic involvement secondary to RA such as vasculitis, pulmonary fibrosis or Felty's syndrome
* History of or current autoimmune or rheumatic disorders, other than RA
* RA functional class 4 or other uncontrolled medical conditions
* History of ongoing, chronic or recurrent infections or recent serious or life-threatening infection
* Presence of any condition that could, in the opinion of the investigator, compromise the individual's ability to participate in the study, such as history of substance abuse, alcoholism, or a psychiatric condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (9):
- United States (9):
  - UC Davis Lawrence J. Ellison, Sacramento, California
  - SeaView Research, Inc., Miami, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Lovelace Scientific Resources, Inc., Venice, Florida
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Justus J. Fiechtner, M.D., P.C., Lansing, Michigan
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Arthritis & Osteoporosis Center of South Texas, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 11 study sites in the United States. The first participant was screened on 26 January 2016. The last study visit occurred on 01 September 2016.
Pre-assignment Details: 58 participants were screened and 42 participants were enrolled.
Period: Overall Study
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 1, Part A: Placebo | Cohort 2, Part A: Tirabrutinib 10 mg BID | Cohort 2, Part A: Placebo | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Started | 8 | 2 | 8 | 2 | 17 | 5
Completed | 8 | 2 | 8 | 2 | 16 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Randomized but Never Treated | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 1, Part A: Placebo | Cohort 2, Part A: Tirabrutinib 10 mg BID | Cohort 2, Part A: Placebo | Part B: Tirabrutinib 20 mg QD | Part B: Placebo | Total
Number analyzed (Participants) | 8 | 2 | 8 | 2 | 16 | 5 | 41
Age, Continuous [Mean (Full Range); unit: years] | 38 [30 to 44] | 37 [29 to 44] | 34 [22 to 45] | 38 [33 to 43] | 55 [38 to 64] | 52 [35 to 64] | 45.5 [22 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 0 | 13 | 4 | 24
  Male | 4 | 1 | 6 | 2 | 3 | 1 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 8 | 2 | 2 | 2 | 24
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 14 | 3 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 4 | 0 | 0 | 1 | 0 | 0 | 5
  Race: White | 4 | 2 | 8 | 1 | 16 | 5 | 36

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Treatment-emergent adverse events (TEAEs) were defined as 1 or both of the following: Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or Any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date up to last dose (maximum: 7 days) plus 30 days
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 2, Part A: Placebo: Placebo to match tirabrutinib 10 mg capsules orally BID (morning and approximately 12 hours later) for 7 days. On Day 7, only morning dose was administered.
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 1, Part A: Placebo | Cohort 2, Part A: Tirabrutinib 10 mg BID | Cohort 2, Part A: Placebo
Number analyzed (Participants) | 8 | 2 | 8 | 2
percentage of participants | 25.0 | 50.0 | 37.5 | 0

2. Primary Outcome: Part A: Percentage of Participants With Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from the predose assessment after the first dose of study drug and within 30 days after last study drug administration. Laboratory abnormalities without clinical significance were not recorded as AEs or serious AEs. Treatment-emergent laboratory abnormalities were graded per Common Terminology Criteria for Adverse Events (CTCAE), version 4.03 where 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = potentially life threatening.
Time Frame: First dose date up to last dose (maximum: 7 days) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1, Part A: Tirabrutinib 20 mg QD: Tirabrutinib 20 mg capsules orally QD in the morning for 1 week.
- Cohort 2, Part A: Tirabrutinib 10 mg BID: Tirabrutinib 10 mg capsules orally BID (morning and approximately 12 hours later) for 7 days. On Day 7, only morning dose was administered.
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 1, Part A: Placebo | Cohort 2, Part A: Tirabrutinib 10 mg BID | Cohort 2, Part A: Placebo
Number analyzed (Participants) | 8 | 2 | 8 | 2
percentage of participants
  Hemoglobin Decreased | 25.0 | 0 | 37.5 | 50.0
  Neutrophils Decreased | 0 | 0 | 0 | 0
  White Blood Cells Decreased | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT) Increased | 25.0 | 0 | 25.0 | 0
  Aspartate Aminotransferase (AST) Increased | 12.5 | 0 | 25.0 | 0
  Alkaline Phosphatase Increased | 0 | 0 | 12.5 | 0
  Amylase | 12.5 | 0 | 0 | 0
  Calcium Increased | 12.5 | 0 | 0 | 0
  Fasting Glucose Increased | 12.5 | 0 | 0 | 0
  Gamma-glutamyl Transferase (GGT) Increased | 25.0 | 0 | 0 | 0
  Glucose Increased | 12.5 | 0 | 0 | 0
  Phosphorus Decreased | 12.5 | 0 | 0 | 0
  Sodium Decreased | 0 | 50.0 | 0 | 0
  Total Cholesterol Increased | 25.0 | 0 | 12.5 | 100.0
  Triglycerides Increased | 25.0 | 0 | 37.5 | 50.0
  Magnesium Increased | 0 | 0 | 0 | 0
  Potassium Decreased | 0 | 0 | 0 | 0

3. Primary Outcome: Part A: Percentage of Participants With 12-Lead Electrocardiogram (ECG) Abnormalities
Time Frame: First dose date up to last dose (maximum: 7 days) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 1, Part A: Placebo | Cohort 2, Part A: Tirabrutinib 10 mg BID | Cohort 2, Part A: Placebo
Number analyzed (Participants) | 8 | 2 | 8 | 2
percentage of participants | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Cmax: Maximum Observed Plasma Concentration of Tirabrutinib
Description: Cmax is maximum observed concentration of drug in plasma.
Time Frame: Cohorts 1 and 2, Day 1: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, and 24 hours postdose; Day 7: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60, 72, 96, and 120 hours postdose
Population: The Pharmacokinetics (PK) Analysis Set included all randomized participants who received at least 1 dose of tirabrutinib and had at least 1 non-missing PK concentration data reported by the PK lab for each respective analyte.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 2, Part A: Tirabrutinib 10 mg BID
Number analyzed (Participants) | 8 | 8
nanogram per milliliter (ng/mL)
  Day 1 | 33.8 (7.94) | 16.2 (4.66)
  Day 7 | 56.4 (11.19) | 32.3 (8.59)

5. Primary Outcome: Part A: Clast: Last Observed Quantifiable Plasma Concentration of Tirabrutinib
Description: Clast is the last observed concentration of drug in plasma.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 2, Part A: Tirabrutinib 10 mg BID
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 | 2.58 (1.366) | 5.22 (1.729)
  Day 7 | 1.50 (0.551) | 2.03 (0.756)

6. Primary Outcome: Part A: Tmax: Time (Observed Time Point) of Cmax of Tirabrutinib
Description: Tmax is the time observed for the Cmax of tirabrutinib.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 2, Part A: Tirabrutinib 10 mg BID
Number analyzed (Participants) | 8 | 8
hours
  Day 1 | 2.00 [1.50 to 4.00] | 3.00 [1.50 to 4.00]
  Day 7 | 2.00 [1.50 to 3.00] | 2.00 [1.50 to 4.00]

7. Primary Outcome: Part A: Tlast: Time (Observed Time Point) of Clast of Tirabrutinib
Description: Tlast is the time observed for the Clast of tirabrutinib.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 2, Part A: Tirabrutinib 10 mg BID
Number analyzed (Participants) | 8 | 8
hours
  Day 1 | 23.92 [12.00 to 23.92] | 11.92 [11.92 to 12.00]
  Day 7 | 30.00 [24.00 to 48.00] | 24.00 [18.00 to 36.00]

8. Primary Outcome: Part A: AUCtau: Area Under the Plasma Concentration (AUC) Versus Time Curve Over the Dosing Interval of Tirabrutinib
Description: AUC is concentration of drug over time (area under the plasma concentration versus time curve).
Time Frame: Cohorts 1 and 2, Day 7: 0 (predose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60, 72, 96, and 120 hours postdose relative to the morning dose
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 2, Part A: Tirabrutinib 10 mg BID
Number analyzed (Participants) | 8 | 8
hours*nanogram per milliliter (h*ng/mL) | 360.5 (97.49) | 195.2 (44.43)

9. Primary Outcome: Part A: AUClast: AUC Versus Time Curve From Time Zero to the Last Quantifiable Concentration of Tirabrutinib
Description: AUC is concentration of drug over time (area under the plasma concentration versus time curve).
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 2, Part A: Tirabrutinib 10 mg BID
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Day 1 | 228.3 (89.96) | 107.1 (27.54)
  Day 7 | 377.8 (119.80) | 245.5 (65.02)

10. Primary Outcome: Part B: Percentage of Participants Who Experienced TEAEs
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs were defined as 1 or both of the following: Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug and/or Any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date up to last dose (maximum: 29 days) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants | 37.5 | 40.0

11. Primary Outcome: Part B: Percentage of Participants With Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from the predose assessment after the first dose of study drug and within 30 days after last study drug administration. Laboratory abnormalities without clinical significance were not recorded as AEs or serious AEs. Treatment-emergent laboratory abnormalities were graded per CTCAE, version 4.03 where 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = potentially life threatening.
Time Frame: First dose date up to last dose (maximum: 29 days) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Hemoglobin Decreased | 6.3 | 0
  Neutrophils Decreased | 6.3 | 0
  White Blood Cells Decreased | 6.3 | 0
  Alanine Aminotransferase (ALT) Increased | 12.5 | 20.0
  Fasting Glucose Increased | 12.5 | 20.0
  Glucose Increased | 12.5 | 20.0
  Magnesium Increased | 18.8 | 0
  Potassium Decreased | 12.5 | 0

12. Primary Outcome: Part B: Percentage of Participants With 12-Lead ECG Abnormalities
Time Frame: First dose date up to last dose (maximum: 29 days) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants | 0 | 0

13. Secondary Outcome: Part A: Change From Baseline in Percent Inhibition of CD63 Basophils at Days 1, 3, 5 and 7
Description: The effect of tirabrutinib on biomarkers was assessed through the CD63 basophil activation test (BAT) FlowCast assay, which was used to measure the percentage of CD63+ basophils and percentage inhibition of CD63 induction relative to baseline. CD63+ % inhibition was calculated as 100 - CD63+ % baseline. Baseline defined as day 1 predose.
Time Frame: Days 1 and 7: Predose and 2, 6, 12, 24 hours postdose; Days 3 and 5: Predose and 2 hours postdose
Population: The Biomarker Analysis Set included all randomized participants who received at least 1 dose of study drug and for whom biomarker data were available.
Measure: Mean (Standard Deviation); unit: percentage of Inhibition
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 1, Part A: Placebo | Cohort 2, Part A: Tirabrutinib 10 mg BID | Cohort 2, Part A: Placebo
Number analyzed (Participants) | 7 | 2 | 8 | 2
percentage of Inhibition
  Day 1, Predose | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Day 1, 2 Hours Postdose | 17.189 (6.8306) | 0.272 (2.3326) | 19.557 (11.0479) | 3.568 (1.4734)
  Day 1, 6 Hours Postdose | 34.966 (15.6436) | 8.779 (9.9101) | 27.506 (16.0744) | 1.782 (6.3117)
  Day 1, 12 Hours Postdose: number analyzed (Participants) | 0 | 0 | 8 | 2
  Day 1, 12 Hours Postdose |  |  | 35.008 (24.1663) | -2.688 (16.7688)
  Day 1, 24 Hours Postdose: number analyzed (Participants) | 7 | 2 | 0 | 0
  Day 1, 24 Hours Postdose | 33.305 (14.9248) | 5.604 (1.2275) |  |
  Day 3, Predose | 47.416 (17.0470) | 0.917 (11.4281) | 83.832 (10.1042) | -11.354 (16.5029)
  Day 3, 2 Hours Postdose | 73.972 (15.1658) | -0.842 (4.6395) | 90.187 (5.6699) | -13.641 (13.0667)
  Day 5, Predose | 55.680 (21.5018) | 2.779 (3.7023) | 83.380 (10.3976) | -2.271 (0.2060)
  Day 5, 2 Hours Postdose | 80.271 (16.8806) | -0.043 (2.3069) | 91.159 (7.4740) | -15.923 (11.5733)
  Day 7, Predose | 56.986 (20.3972) | 5.234 (0.8757) | 80.024 (11.0371) | 6.271 (7.9790)
  Day 7, 2 Hours Postdose | 79.910 (15.3155) | -2.831 (0.7358) | 88.032 (7.8750) | -0.978 (9.9380)
  Day 7, 6 Hours Postdose | 88.102 (11.6072) | -1.320 (8.1776) | 89.681 (7.0909) | -2.645 (6.3382)
  Day 7, 12 Hours Postdose: number analyzed (Participants) | 0 | 0 | 8 | 2
  Day 7, 12 Hours Postdose |  |  | 80.640 (10.0574) | -10.062 (13.2554)
  Day 7, 24 Hours Postdose: number analyzed (Participants) | 7 | 2 | 0 | 0
  Day 7, 24 Hours Postdose | 52.017 (17.5829) | -0.046 (0.6432) |  |

14. Secondary Outcome: Part A: Change From Baseline in Percent Bruton's Tyrosine Kinase (BTK) Occupancy at Days 1, 3, 5 and 7
Description: BTK occupancy was assessed with the BTK occupancy assay, which was used to measure undetectable free BTK, normalized free BTK, normalized free BTK adjusted to baseline, and percentage BTK occupancy adjusted to baseline. % BTK occupancy adjusted was calculated as 100 * (1 - normalized free BTK adjusted to baseline). Normalized free BTK was calculated as Free BTK / Total BTK. Baseline defined as day 1 predose.
Time Frame: Day 1: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24 hours postdose; Days 3 and 5: Predose and 2 hours postdose; Day 7: Predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 60, 72, 96, 120 hours postdose
Population: Participants in the Biomarker Analysis Set were analyzed. All of the baseline samples collected for BTK occupancy assay in Part A Cohort 2 were compromised and therefore not evaluable.
Measure: Mean (Standard Deviation); unit: percentage of BTK occupancy
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 1, Part A: Placebo
Number analyzed (Participants) | 7 | 2
percentage of BTK occupancy
  Day 1, Predose | 0 (0) | 0 (0)
  Day 1, 0.5 Hour Postdose | -2.765 (14.6036) | -4.686 (1.8358)
  Day 1, 1 Hour Postdose | 11.635 (17.8025) | -11.927 (8.4893)
  Day 1, 2 Hours Postdose | 55.250 (10.0230) | -8.959 (16.7122)
  Day 1, 3 Hours Postdose | 62.719 (7.7060) | -9.810 (18.8212)
  Day 1, 4 Hours Postdose | 66.790 (7.9494) | -16.597 (25.0492)
  Day 1, 6 Hours Postdose | 71.936 (8.3606) | -6.014 (19.5348)
  Day 1, 8 Hours Postdose | 75.350 (11.5216) | -16.584 (17.8202)
  Day 1, 12 Hours Postdose | 77.411 (8.6928) | 6.170 (12.7312)
  Day 1, 18 Hours Postdose | 81.187 (8.8687) | -2.261 (27.3338)
  Day 1, 24 Hours Postdose | 72.691 (10.8289) | -28.029 (10.1821)
  Day 3, Predose | 84.010 (8.4919) | -19.564 (20.3282)
  Day 3, 2 Hours Postdose | 90.606 (6.1066) | -35.206 (25.2258)
  Day 5, Predose | 70.841 (43.0596) | 25.095 (99.0827)
  Day 5, 2 Hours Postdose | 93.128 (4.0582) | -25.646 (17.6912)
  Day 7, Predose | 86.936 (6.4745) | -22.662 (23.6252)
  Day 7, 0.5 Hours Postdose | 87.013 (5.2426) | -23.284 (9.9539)
  Day 7, 1 Hour Postdose | 86.274 (6.0720) | -12.230 (6.6727)
  Day 7, 2 Hours Postdose | 92.651 (3.4603) | -34.573 (17.9620)
  Day 7, 3 Hours Postdose | 92.983 (2.1906) | -32.920 (20.1029)
  Day 7, 4 Hours Postdose | 90.070 (7.4086) | -37.253 (16.2208)
  Day 7, 6 Hours Postdose | 91.591 (7.7733) | -39.632 (13.1749)
  Day 7, 8 Hours Postdose | 92.789 (3.2221) | -31.144 (20.1974)
  Day 7, 12 Hours Postdose | 91.251 (6.0300) | -33.947 (16.3475)
  Day 7, 18 Hours Postdose | 85.209 (5.0694) | -34.408 (12.5471)
  Day 7, 24 Hours Postdose | 86.256 (6.5648) | -42.577 (17.2138)
  Day 7, 36 Hours Postdose | 71.963 (10.5550) | -43.574 (8.4952)
  Day 7, 48 Hours Postdose | 64.763 (14.3072) | -46.249 (24.2785)
  Day 7, 60 Hours Postdose | 57.431 (9.0638) | -15.465 (9.4556)
  Day 7, 72 Hours Postdose | 46.218 (14.3155) | -49.093 (21.4447)
  Day 7, 96 Hours Postdose | 24.922 (6.8700) | -41.721 (32.0255)
  Day 7, 120 Hours Postdose | 15.285 (9.4140) | -48.863 (20.7533)

15. Secondary Outcome: Part B: Change From Baseline in Disease Activity Score for 28 Joint Counts (DAS28) Using C-Reactive Protein (CRP) at Weeks 2, 4 and Posttreatment Week 4
Description: DAS28 score was used to measure the participant's disease activity or assessments of rheumatoid arthritis (RA) calculated using the tender joint counts (TJC) (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (PtGA) (visual analog scale: 0 = no disease activity to 100 = maximum disease activity) and CRP for a total possible score of 2 to 10. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set (who were randomized into the study and received at least 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
score on a scale
  Baseline | 4.54 (1.728) | 5.12 (1.576)
  Change from Baseline at Week 2 | -0.35 (0.821) | -0.28 (0.977)
  Change from Baseline at Week 4 | -0.45 (1.097) | -0.11 (0.612)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -0.41 (1.208) | -0.05 (0.782)

16. Secondary Outcome: Part B: Change From Baseline in Individual American College of Rheumatology (ACR) Component: Tender Joint Count (TJC) Based on 68 Joints (TJC68) at Weeks 2, 4 and Posttreatment Week 4
Description: ACR TJC was an assessment of 68 joints. At each study visit, a joint evaluator assessed whether a particular joint was "tender" where presence of tenderness was scored as "1" and the absence of tenderness was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons. It was derived as the sum of all tender joints. The range for TJC68 was 0 to 68, with a higher score indicating a greater degree of tenderness. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
tender joint count
  Baseline | 18.20 (14.454) | 21.70 (12.656)
  Change from Baselline at Week 2 | -2.57 (6.666) | -1.17 (7.980)
  Change from Baselline at Week 4: number analyzed (Participants) | 16 | 4
  Change from Baselline at Week 4 | -6.69 (8.432) | 0.01 (0.829)
  Change from Baselline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baselline at Posttreatment Week 4 | -3.13 (9.968) | 1.11 (12.638)

17. Secondary Outcome: Part B: Change From Baseline in Individual ACR Component: Swollen Joint Count (SJC) Based on 66 Joints (SJC66) at Weeks 2, 4 and Posttreatment Week 4
Description: ACR SJC was an assessment of 66 joints. At each study visit, a joint evaluator assessed whether a particular joint was swollen where presence of swelling was scored as "1" and the absence of swelling was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons. It was derived as the sum of all swollen joints. The range for SJC66 was 0 to 66, with a higher score indicating a greater degree of swelling. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
swollen joint count
  Baseline | 12.70 (10.944) | 12.04 (12.488)
  Change from Baseline at Week 2 | -4.13 (6.446) | -2.58 (9.910)
  Change from Baseline at Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Week 4 | -4.82 (7.586) | -2.23 (6.048)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -3.07 (5.272) | 1.53 (3.035)

18. Secondary Outcome: Part B: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 2, 4 and Posttreatment Week 4
Description: SDAI is a composite measure that sums the TJC based on 28 joints (TJC28), SJC based on 28 joints (SJC28), PtGA, Physician's Global Assessment of Disease Activity (PhGA), and the CRP (in mg/dL). PtGA and PhGA assessed using Visual Analogue Scale (VAS) on a scale of 0-100 [0 indicating no disease activity and 100 indicating maximum disease activity]. SDAI total score range: 0 to 86. SDAI <= 3.3 indicates disease remission and SDAI > 26 = high disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
score on a scale
  Baseline | 30.19 (20.283) | 33.20 (19.061)
  Change from Baseline at Week 2 | -4.49 (11.786) | -5.20 (14.035)
  Change from Baseline at Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Week 4 | -6.84 (14.016) | -1.69 (5.439)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -4.82 (14.349) | -1.16 (12.293)

19. Secondary Outcome: Part B: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 2, 4 and Posttreatment Week 4
Description: CDAI is a composite measure that sums the TJC28, SJC28, PtGA, and PhGA. PtGA and PhGA assessed using VAS on a scale of 0-100 [0 indicating no disease activity and 100 indicating maximum disease activity]. CDAI total score range: 0 to 76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity, and > 22 = high disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
score on a scale
  Baseline | 29.63 (19.994) | 31.96 (18.622)
  Change from Baseline at Week 2 | -4.44 (11.748) | -5.32 (13.264)
  Change from Baseline at Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Week 4 | -6.80 (13.925) | -2.02 (5.206)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -4.73 (14.180) | -1.74 (11.562)

20. Secondary Outcome: Part B: Change From Baseline in Individual ACR Component: Patient's Global Assessment of Disease Activity (PtGA) at Weeks 2, 4 and Posttreatment Week 4
Description: PtGA was assessed by the participant using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A horizontal visual analog scale was used to provide the patient's overall assessment of how the arthritis is doing. A mark was placed on the horizontal line to assess the current arthritis disease activity. The lowest mark indicated 'no arthritis activity', and the highest mark indicated 'extremely active arthritis'. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
score on a scale
  Baseline | 42 (27.4) | 63 (30.5)
  Change from Baseline at Week 2 | -10 (20.7) | -6 (17.6)
  Change from Baseline at Week 4 | -10 (22.1) | -10 (16.7)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -4 (22.2) | -9 (17.8)

21. Secondary Outcome: Part B: Change From Baseline in Individual ACR Component: Physician's Global Assessment of Disease Activity (PhGA) at Weeks 2, 4 and Posttreatment Week 4
Description: PhGA was assessed by the physician using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A horizontal visual analog scale was used to measure the physician's assessment of the patient's current disease activity. A mark was placed on the horizontal line to assess the disease activity (independent of the participant's self-assessment). The lowest mark indicated 'no disease activity', and the highest mark indicated 'maximum disease activity'. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
score on a scale
  Baseline | 39 (27.4) | 49 (15.5)
  Change from Baseline at Week 2 | -3 (23.5) | -16 (13.4)
  Change from Baseline at Week 4 | -8 (20.3) | 5 (14.9)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -4 (22.7) | -3 (17.7)

22. Secondary Outcome: Part B: Change From Baseline in Individual ACR Component: Patient's Global Assessment of Pain at Weeks 2, 4 and Posttreatment Week 4
Description: The participant assessed their pain severity using a VAS on a scale of 0 (no pain) to 100 (severe pain). A horizontal visual analog scale was used to assess the patient's current level of pain. A mark was placed on the horizontal line to assess the severity of pain. The lowest mark indicated 'no pain', and the highest mark indicated 'unbearable pain'. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
score on a scale
  Baseline | 39 (28.6) | 59 (28.9)
  Change from Baseline at Week 2 | -5 (26.2) | -6 (15.7)
  Change from Baseline at Week 4 | -9 (24.6) | -13 (16.2)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -2 (22.9) | -11 (24.9)

23. Secondary Outcome: Part B: Change From Baseline in the Health Assessment Questionnaire Disability Subscales (HAQ-DI) Score at Weeks 2, 4 and Posttreatment Week 4
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually administered by the participant. Responses in each functional category were collected as 0-3 [0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
score on a scale
  Baseline | 1.063 (0.7130) | 1.650 (0.7776)
  Change from Baseline at Week 2 | -0.203 (0.5242) | -0.150 (0.2054)
  Change from Baseline at Week 4 | -0.234 (0.4492) | -0.100 (0.3687)
  Change from Baseline at Posttreatment Week 4: number analyzed (Participants) | 16 | 4
  Change from Baseline at Posttreatment Week 4 | -0.156 (0.3550) | 0.094 (0.1197)

24. Secondary Outcome: Part B: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement (ACR20) Response at Weeks 2, 4 and Posttreatment Week 4
Description: ACR20 response is achieved when the participant has: ≥ 20% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PhGA and PtGA assessed using VAS on a scale of 0-100 (0 and 100 indicating no disease activity and maximum disease activity); patient's pain assessment using VAS on a scale of 0-100 (0 indicating no pain and 100 indicating unbearable pain); HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 (0 and 3 indicating without difficulty and unable to do); high-sensitivity CRP (hsCRP).
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Week 2 | 6.3 | 20.0
  Week 4 | 18.8 | 0
  Posttreatment Week 4 | 12.5 | 0

25. Secondary Outcome: Part B: Percentage of Participants Who Achieved ACR 70% Improvement (ACR70) Response at Weeks 2, 4 and Posttreatment Week 4
Description: ACR70 response is achieved when the participant has: ≥ 70% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PhGA and PtGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; patient's pain assessment using VAS on a scale of 0-100 [0 indicating no pain and 100 indicating unbearable pain]; HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  At Week 2 | 0 | 0
  At Week 4 | 6.3 | 0
  At Posttreatment Week 4 | 0 | 0

26. Secondary Outcome: Part B: Hybrid ACR Improvement Response at Weeks 2, 4 and Posttreatment Week 4
Description: Hybrid ACR evaluates the improvement in active RA by combining elements of the ACR20, ACR50, and ACR70 with a continuous score of the mean change in core set measures. The percentage improvement from baseline was computed in each of the components of the ACR. The average percent improvement was calculated and used with the participant's ACR20, ACR50, and ACR70 status to compute the hybrid ACR response, with a positive change indicating improvement.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percent improvement
  At Week 2: number analyzed (Participants) | 15 | 5
  At Week 2 | 1.51 (30.687) | 4.41 (25.410)
  At Week 4: number analyzed (Participants) | 16 | 4
  At Week 4 | 3.29 (36.098) | -4.06 (14.459)
  At Posttreatment Week 4: number analyzed (Participants) | 15 | 4
  At Posttreatment Week 4 | 0.44 (34.589) | -7.65 (20.606)

27. Secondary Outcome: Part B: Percentage of Participants Who Achieved Remission as Measured by DAS28-CRP at Weeks 2, 4 and Posttreatment Week 4
Description: Clinical remission is defined as DAS28-CRP < 2.6. DAS28 score was used to measure the participant's disease activity or assessments of RA calculated using the TJC28, SJC28, PtGA (VAS: 0 = no disease activity to 100 = maximum disease activity) and CRP for a total possible score of 2 to 10. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Week 2: Remission based on DAS28-CRP (< 2.6) | 12.5 | 0
  Week 4: Remission based on DAS28-CRP (< 2.6) | 12.5 | 0
  Post Week 4: Remission based on DAS28-CRP (< 2.6) | 25.0 | 0

28. Secondary Outcome: Part B: Percentage of Participants Who Achieved Low Disease Activity Response as Measured by DAS28-CRP at Weeks 2, 4 and Posttreatment Week 4
Description: Low disease activity is defined as DAS28-CRP ≤ 3.2. DAS28 score was used to measure the participant's disease activity or assessments of RA calculated using the TJC28, SJC28, PtGA (VAS: 0 = no disease activity to 100 = maximum disease activity) and CRP for a total possible score of 2 to 10. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Week 2: Low Disease Activity on DAS28-CRP (<= 3.2) | 18.8 | 20.0
  Week 4: Low Disease Activity on DAS28-CRP (<= 3.2) | 12.5 | 20.0
  Post Week4: Low Disease Activity DAS28-CRP (<=3.2) | 37.5 | 0

29. Secondary Outcome: Part B: Percentage of Participants Who Achieved Remission as Measured by CDAI at Weeks 2, 4 and Posttreatment Week 4
Description: Clinical remission is defined as CDAI ≤ 2.8. CDAI is a composite measure that sums the TJC28, SJC28, PtGA, and PhGA. PtGA and PhGA assessed using VAS on a scale of 0-100 [0 indicating no disease activity and 100 indicating maximum disease activity]. CDAI total score range: 0 to 76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity, and > 22 = high disease activity. A negative change from baseline indicates improvement.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Week 2: Remission based on CDAI (<= 2.8) | 12.5 | 0
  Week 4: Remission based on CDAI (<= 2.8) | 6.3 | 0
  Post Week 4: Remission based on CDAI (<= 2.8) | 6.3 | 0

30. Secondary Outcome: Part B: Percentage of Participants Who Achieved Low Disease Activity Response as Measured by CDAI at Weeks 2, 4 and Posttreatment Week 4
Description: Low disease activity is defined as CDAI ≤ 10. CDAI is a composite measure that sums the TJC28, SJC28, PtGA, and PhGA. PtGA and PhGA assessed using VAS on a scale of 0-100 [0 indicating no disease activity and 100 indicating maximum disease activity]. CDAI total score range: 0 to 76. CDAI <= 2.8 indicates disease remission, > 2.8 to 10 = low disease activity, > 10 to 22 = moderate disease activity, and > 22 = high disease activity. A negative change from baseline indicates improvement.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Week 2: Low Disease Activity based on CDAI (<= 10) | 18.8 | 20.0
  Week 4: Low Disease Activity based on CDAI (<= 10) | 18.8 | 20.0
  Post Week 4: Low Disease Activity on CDAI (<= 10) | 31.3 | 20.0

31. Secondary Outcome: Part B: Percentage of Participants Who Achieved Remission as Measured by SDAI at Weeks 2, 4 and Posttreatment Week 4
Description: Clinical remission is defined as SDAI ≤ 3.3. SDAI is a composite measure that sums the TJC28, SJC28, PtGA, PhGA, and the CRP (in mg/dL). PtGA and PhGA assessed using VAS on a scale of 0-100 [0 indicating no disease activity and 100 indicating maximum disease activity]. SDAI total score range: 0 to 86. SDAI <= 3.3 indicates disease remission and SDAI > 26 = high disease activity. A negative change from baseline indicates improvement.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Week 2: Remission based on SDAI (<= 3.3) | 12.5 | 0
  Week 4: Remission based on SDAI (<= 3.3) | 6.3 | 0
  Post Week 4: Remission based on SDAI (<= 3.3) | 6.3 | 0

32. Secondary Outcome: Part B: Percentage of Participants Who Achieved Low Disease Activity Response as Measured by SDAI at Weeks 2, 4 and Posttreatment Week 4
Description: Low disease activity is defined as SDAI ≤ 11. SDAI is a composite measure that sums the TJC28, SJC28, PtGA, PhGA, and the CRP (in mg/dL). PtGA and PhGA assessed using VAS on a scale of 0-100 [0 indicating no disease activity and 100 indicating maximum disease activity]. SDAI total score range: 0 to 86. SDAI <= 3.3 indicates disease remission and SDAI > 26 = high disease activity. A negative change from baseline indicates improvement.
Time Frame: Weeks 2, 4 and Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Tirabrutinib 20 mg QD | Part B: Placebo
Number analyzed (Participants) | 16 | 5
percentage of participants
  Week 2: Low Disease Activity based on SDAI (<= 11) | 25.0 | 20.0
  Week 4: Low Disease Activity based on SDAI (<= 11) | 18.8 | 20.0
  Post Week 4: Low Disease Activity on SDAI (<= 11) | 37.5 | 20.0

ADVERSE EVENTS:
Time Frame: Adverse Events: Part A: First dose date up to last dose (maximum: 7 days) plus 30 days; Part B: First dose date up to last dose (maximum: 29 days) plus 30 days; All-Cause Mortality: First dose date up to approximately 7 months
Description: Participants in the Safety Analysis Set were analyzed.
Groups:
- All Placebo: Cohort 1, Part A: Placebo to match tirabrutinib capsules orally QD in the morning for 1 week; Cohort 2, Part A: Placebo to match tirabrutinib capsules orally BID (morning and approximately 12 hours later) for 7 days. On Day 7, only morning dose was administered. Part B, Placebo to match tirabrutinib capsules orally QD for 4 weeks.
Arm/Group | Cohort 1, Part A: Tirabrutinib 20 mg QD | Cohort 2, Part A: Tirabrutinib 10 mg BID | Part B: Tirabrutinib 20 mg QD | All Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/16 | 0/9
Other Adverse Events (participants affected / at risk) | 2/8 | 3/8 | 6/16 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Part A: Tirabrutinib 20 mg QD (N=8) | Cohort 2, Part A: Tirabrutinib 10 mg BID (N=8) | Part B: Tirabrutinib 20 mg QD (N=16) | All Placebo (N=9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Extravasation (General disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years